CLINICAL TRIAL: NCT06777238
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Chinese Subjects With Type 2 Diabetes Mellitus and Poor Blood Glucose Control by Diet and Exercise
Brief Title: A Phase III Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Subjects With Type 2 Diabetes Mellitus and Poor Blood Glucose Control by Diet and Exercise
Acronym: Optimum 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZR18-T2DM-301
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: GLP-1RA
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GZR18 Dose1 (Experimental): Participants will receive GZR18 subcutaneously (SC).
  Interventions: Drug: GZR18
- GZR18 Dose 2 (Experimental): Participants will receive GZR18 subcutaneously (SC).
  Interventions: Drug: GZR18
- placebo group (Placebo Comparator): Participants will receive placebo subcutaneously (SC).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GZR18 — Administered SC
  Arms: GZR18 Dose 2; GZR18 Dose1
Drug: Placebo — Administered SC
  Arms: placebo group

SUMMARY:
The main purpose of this study is to investigate the Efficacy and Safety of GZR18 Injection in Chinese Subjects with Type 2 Diabetes Mellitus and Poor Blood Glucose Control by Diet and Exercise

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (as of the date of signing the Informed Consent Form (ICF)), male or female.
2. T2DM is diagnosed for at least 8 weeks according to the diagnostic criteria of diabetes mellitus issued by the World Health Organization (WHO) in 1999 and the supplementary diagnostic criteria of WHO in 2011 (HbA1c diagnosis is recommended).
3. No birth plan from the signing of ICF to 8 weeks after the last dose, willingness to use effective methods of contraception, and no plan for sperm donation. Females of childbearing potential must not be lactating and must have negative results of pregnancy tests at screening and baseline.
4. Fully understand the purpose, nature, methods, and possible adverse drug reactions (ADRs) of the study, be able to communicate well with the investigator, can understand and comply with the requirements specified in this study, can maintain a regular diet and exercise lifestyle during the study, and voluntarily sign the ICF to enter the study.

   -

Exclusion Criteria:

1. Poor compliance during the run-in period as assessed by the investigator.
2. Known or suspected to be allergic to GLP-1R agonists or their excipients, or have contraindications to their use.

（3)Systolic blood pressure (SBP) ≥ 160 mmHg or diastolic blood pressure (DBP) ≥ 100 mmHg at screening or before randomization (concomitant antihypertensive drugs are allowed).

（4）Have the following cardiovascular and cerebrovascular diseases within 6 months before screening: Decompensated cardiac insufficiency (New York Heart Association NYHA Class III or IV), angina unstable or myocardial infarction, history of heart valve replacement surgery, coronary artery bypass grafting or other invasive cardiovascular surgery including percutaneous coronary intervention, ischemic or hemorrhagic stroke (excluding lacunar infarction), or transient ischemic attack.

（5）History or relevant family history of medullary thyroid cancer, multiple endocrine neoplasia (MEN) 2A or 2B before screening.

（6）History of malignant tumors before screening (excluding adequately treated or resected non-metastatic basal or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer in situ) or the presence of underlying malignancy at screening.

（7）Participated in any drug clinical study (received non-placebo medication during the study) within a period of time before randomization (90 days or 5 half-lives of the previous IMP, whichever is longer), or plan to participate in another clinical study before completing all scheduled assessments in this clinical study.

（8）Subjects with any other factors that may affect the efficacy or safety evaluation of this study as judged by the investigator.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Baseline, Week 44
  Change in HbA1c

SECONDARY OUTCOMES:
Change in weight（Kg）. | Baseline, Week 44
Change in BMI（kg/m2）. | Baseline, Week 44
Change in waist circumference(cm). | Baseline, Week 44
Change in hip circumference(cm). | Baseline, Week 44

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: No